CLINICAL TRIAL: NCT00334373
Title: Post Conditioning in PCI for Acute ST Elevation Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Foothills Interventional Cardiology Research Group (Unknown)
Responsible Party: Principal Investigator, Todd Anderson, Director Libin Cardiovascular Institute, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ethics ID E-20039
Record Dates: First submitted 2006-06-06; First posted 2006-06-07 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Myocardial Infarction
Keywords: Myocardial infarction; Magnetic Resonance Imaging; Coronary Angioplasty
MeSH Terms: conditions — Myocardial Infarction | interventions — Ischemic Postconditioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Post conditioning (Experimental): Balloon inflations-deflations
  Interventions: Procedure: Post conditioning
- Standard care (Placebo Comparator): No balloon inflations
  Interventions: Procedure: Post conditioning

INTERVENTIONS:
Procedure: Post conditioning — 4 cycles of balloon inflation /deflation (post-conditioning) within first minute of opening up artery in primary PCI for STEMI vs usual balloon inflation sequence

SUMMARY:
The purpose of this trial is to compare post-conditioning to standard angioplasty (50/50 chance) in patients who present with an acute heart attack and are taken directly for an angioplasty procedure. Post conditioning is a procedure that involves balloon inflation followed by deflation in a series of cycles that appears to show (based on early data) that it can decrease the amount of damage to the heart muscle as compared to standard angioplasty procedures.

Hypothesis: For Subjects undergoing direct PCI for STEMI, post conditioning with cycles of balloon inflation/deflation within the first minute following the re-establishment of coronary blood blow, will decrease the amount of irreversible myocardial damage assessed by delayed enhancement contrast CMR.

DETAILED DESCRIPTION:
In patients who suffer a myocardial infarction, the blood flow usually ceases due to plaque rupture leading to thrombus formation and vessel occlusion. The resultant entity is known as ST Elevation segment myocardial infarction (STEMI) and is a significant health issue in industrialized countries. There are over 50,000 STEMI's every year in Canada and up to 10% of these patients die in hospital and another 10% die within the first year after their heart attack. The more common problem however is not death, but irreparable damage to the left ventricle leading to LV dysfunction and subsequent heart failure and arrythmias. Re-establishing blood flow promptly by administering plasminogen activators (lytics) or mechanically by performing angioplasty is possible and has lowered the mortality rate dramatically.

Although reperfusion is necessary, it gives rise to an entity known as ischemia-reperfusion where acutely re-establishing blood flow and oxygen levels of the heart has detrimental effects. Clinically this is manifested as no-reflow that causes subsequent damage to the left ventricle and decreases the beneficial affect of early reperfusion by PCI. The ischemia-reperfusion effect sets off a molecular cascade of events involving unfavorable interaction between neutrophils, platelets and endothelium, that is fairly well identified. Efforts to pharmacologically block this effect have not proven to be particularly effective.

Post conditioning follows from a concept of pre-conditioning in animals that showed a decrease in myocardial infarct size. Pre-conditioning is not useful as it requires to be performed prior to the development of ischemia/injury. Post conditioning in preliminary studies with animals and one small study in humans have shown promising results for decrease in infarct size. Post conditioning is a procedure of gradual conditioning in which the artery is opened and closed in cycles with inflation/deflation of the culprit artery followed immediately by standard PCI and placement of stent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* ST elevation of >/= 2mm in 3 consecutive anterior leads or >/= to 2 mm in leads II, III and AVF with total 8 mm ST shift (ST depression of 1 mm in ant or lat leads)

Exclusion Criteria:

* Cardiogenic shock or severe heart failure
* Inability to undergo CMR (metallic objects or claustrophobia)
* Previous MI
* TIMI 2-3 flow in target artery
* Collaterals to infarct related artery > Rentrop grade 1
* Inability to undertake successful PCI at time of angio
* Significant LM disease or requiring CABG during hospital stay
* Inability to proceed with post conditioning within 1 minute of establishing blood flow in culprit artery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Infarct size as measured by: salvage index = total area at risk - infarct size/total area at risk | 3-5 days post MI

SECONDARY OUTCOMES:
Corrected TIMI frame count (cTFC) | Immediately post PCI
Myocardial blush score | Immediately post PCI
CK release (under the curve) | 1st 48 hours post MI
ST segment resolution by 48 hrs compared with admission | 1st 48 hours post MI
MRI infarct size | 3-5 days and 6 months
MRI maximal transmural extent of irreversible injury | 3-5 days and 6 months
CMR regional end-systolic wall stress | 3-5 days and 6 months
CMR Myocardial perfusion | 3-5 days and 6 months
CMR Myocardial oxygenation | 3-5 days and 6 months
Peripheral endothelial function testing (brachial u/s and pulse arterial tonometry) in hospital | 3-5 days post MI
CMR quantification of volume of no-reflow | 3-5 days and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mouhieddin Traboulsi, MD, Study Director — University of Calgary, sub-investigator; Matthias Friedrich, MD, Study Chair — Sub-investigator, Stephenson CMR Centre, FMC; 1403-29th St NW, Calgary; T2N 2T9
Locations (1):
- Foothills Medical Centre, Calgary, Alberta, Canada